CLINICAL TRIAL: NCT03799536
Title: Open-label, Randomized, Crossover, Two-period, Two-sequence Bioequivalence Study of Sotalol, Tablets, 160 mg (Pharmtechnology LLC, Belarus), and Sotalex®, Tablets, 160 mg (BRISTOL-MYERS SQUIBB GmbH & Co. KGaA, Germany), in Healthy Volunteers Under Fasting Condition
Brief Title: Bioequivalence Study of Sotalol, Tablets, 160 mg (Pharmtechnology LLC, Belarus), and Sotalex ®, Tablets, 160 mg (Bristol-Myers Squibb GmbH & Co. KGaA, Germany), in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: National Anti-Doping Labaratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BE-SOTL-160- 2018
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-01

CONDITIONS: Bioequivalence
Keywords: Bioequivalence; Sotalol; Sotalex
MeSH Terms: interventions — Sotalol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The subjects and the investigator will not be blinded towards the identity of the study products. However, analysts will be blinded towards identity of the study products administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental): Subjects assigned to sequence AB will receive a single 160 mg dose of the test product Sotalol (1 x 160 mg tablet) marked as A in the sequence in the period 1 and a single 160 mg dose of the reference product Sotalex (1 x 160 mg tablet) marked as B in the sequence in the period 2 . These treatments will be administered orally with approximately 200 mL of water at ambient temperature, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Sotalol
- Sequence BA (Active Comparator): Subjects assigned to sequence BA will receive a single 160 mg dose of the reference product Sotalex (1 x 160 mg tablet) marked as B in the sequence in the period 1 and a single 160 mg dose of the test product Sotalol (1 x 160 mg tablet) marked as A in the sequence in the period 2 . These treatments will be administered orally with approximately 200 mL of water at ambient temperature, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Sotalex

INTERVENTIONS:
Drug: Sotalol — Sotalol, Tablets,160 mg, manufactured by Pharmtechnology LLC, Belarus
  Other Names: the test product
  Arms: Sequence AB
Drug: Sotalex — Sotalex, Tablets,160 mg, manufactured by Bristol-Myers Squibb GmbH & Co. KGaA, Germany
  Other Names: the reference product
  Arms: Sequence BA

SUMMARY:
This is an open-label, randomized, single-center, single-dose, two-treatment, two-sequence, two-period, crossover, comparative study, where each subject was randomly assigned to the reference or the test formulation in each period of the study (sequences RT or TR), in order to evaluate if both formulations are bioequivalent.The study was conducted in multiple groups.

DETAILED DESCRIPTION:
The objective of this study is to establish if two formulations of sotalol are bioequivalent. The test formulation is Sotalol Tablets, 160 mg (Pharmtechnology LLC, Belarus). The reference formulation is Sotalex®, Tablets, 160 mg (Bristol-Myers Squibb GmbH & Co. KGaA, Germany). 36 healthy adult volunteers of both genders with age ranging from 18 to 55 years old will receive a single tablet (160 mg of sotalol) of the test and the reference products with 200 ml of water after an overnight fast of at least 10 hours, according to the pre-defined randomization list. In the first period, 18 subjects will receive the test product and 18 subjects the reference product.In the second period subjects will receive the products in the opposite order. Subjects will fast 4 hours after administration of the study drugs during each study period. Standardized meals will be provided in each study period. Water will not be accessible to the subjects 1 hour prior to administration of the study drugs and 2 hours after administration of the study drugs in each period. In each period blood samples were collected before dosing and 0,5 ; 1; 1,5; 2 ; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing (total number: 19). The washout period will be 14 days. A validated HPLC/MS/MS method will be used to determine plasma concentrations of analyte (sotalol). ANOVA will be performed on log transformed pharmacokinetic parameters Cmax, AUC0-t and 90% confidence interval will be constructed for the ratio of geometric least square means of the test and the reference products, obtained from the log-transformed data. Bioequivalence will be concluded if the ratio estimate as well as its 90% confidence interval for the analyte, both falls within the acceptable range of 80.00% to 125.00% for Cmax and AUC0-t.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men or women aged between 18 to 55 years
* Body mass index 18.5-30 kg/m²
* Subjects who have no signs of disease during the screening, and whose screening is conducted within 21 days after the registration in the trial
* Subjects whose laboratory blood and urine values are within the normal range orof deviations are considered by researchers to be clinically insignificant
* Non-smokers or ex-smokers (defined as completely quitting smoking for at least three months prior to being included in the test)
* No known history of alcohol abuse
* No known history of abuse of drugs (benzodiazepines, opioids, cocaine, barbiturates, amphetamine, etc.)
* Willingness to comply with the protocol requirements regarding the restriction of the consumption of products containing xanthine (coffee, tea, chocolate, cola, etc.) for at least 48 hours and products containing tobacco, alcohol-containing products and beverages, grapefruit and/or its juice, food containing poppy at least 72 hours prior taking the investigational medicinal products and over the course of the study, as well as requirements regarding the intake of food, fluids and physical activity imposed by the study
* Healthy subject according to medical history, physical examination and assessment of basic vital signs
* No significant abnormalities on 12-lead ECG
* No significant abnormalities on the chest x-ray obtained within 12 months prior the start of the study
* Consent of women of childbearing age and male participants to use medically confirmed barrier methods of contraception (from the date of screening to the completion of the study), or surgical sterilization in history, or women in postmenopause (at least 24 months) or hysterectomy in history . If women use hormonal contraceptives,they should stop them at least 60 days prior the planned beginning of the study
* The subject's voluntary willingness to provide written informed consent
* The ability, at disceretion of the researcher, to follow all the requirements of the protocol
* The ability, at judgment of the researcher, to follow all the requirements of the protocol

Exclusion Criteria:

* Known history of allergy
* Known contraindications to the use of investigational products or hypersensitivity to the active substance or components of drugs
* Use of drugs with enzymatic-modifying activity, within 28 days prior the beginning of the study
* Use any over-the-counter or prescription drugs (including vitamins, minerals, herbal remedies, and dietary supplements) within 14 days prior the administration of investigational products and over the course of the study
* Intense physical exercises within 24 hours prior to the administration of investigational products
* Any medical or surgical interventions that can disrupt the function of the hematopoietic system, the gastrointestinal tract (with the exception of appendectomy), the liver, urinary system and other body systems
* Any chronic diseases or conditions of the urinary, cardiovascular, neuroendocrine, immune, central nervous systems, hematopoietic system, gastrointestinal tract, liver, organs of vision and other systems of the body and diabetes in medical history, mental illness in an active phase or the history
* The presence of any hereditary disease
* Participation in any clinical trials within 90 days prior the beginning of the current clincial study
* Oncological diseaes in medical history
* Any blood donation within 90 days prior the beginning of the current clincial study
* Acute infectious diseases within 28 days prior the beginning of the current clincial study as well as positive testing for HIV, hepatitis B and C, and syphilis
* Positive test for alcohol
* Positive urinary screen test for drugs of abuse
* Swallowing problems in mediical history
* Positive urinary pregnancy test
* Breast-feeding
* Known history of venous access difficulties
* Vegetarian diet
* Sitting systolic blood pressure < 110 mm Hg or > 140 mm Hg and/or sitting diastolic blood pressure < 70 mm Hg or > 90 mm Hg.Heart rate <50 or >100 beats per minute at screening check-in
* Values of the standard laboratory and instrumental tests outside of normal limits and are judged as clinically significant by investigators or require additional examination and interpretation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-11 (Actual)

PRIMARY OUTCOMES:
Cmax of sotalol for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0,5; 1; 1,5; 2; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing
  Maximum concentration in plasma among observed concentrations at pre-specified time points
AUC0-t of sotalol for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0,5; 1; 1,5; 2; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to the last measured concentration

SECONDARY OUTCOMES:
AUC0-∞ of sotalol for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0,5; 1; 1,5; 2; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing
  Area under the plasma concentration versus time curve from time 0 to to infinite time
Tmax of sotalol for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0,5; 1; 1,5; 2; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing
  Time to maximum measured plasma concentration
T1/2 of sotalol for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0,5; 1; 1,5; 2; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing
  Elimination or terminal half-life
Kel of sotalol for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0,5; 1; 1,5; 2; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing
  Elimination rate constant
AUCresid of sotalol for the test and the reference products | Time points: 0,00 (within 30 minutes before dosing) and 0,5; 1; 1,5; 2; 2,5; 3; 3,5; 4; 4,5; 5; 6; 8; 10; 12; 16; 24; 36; 48; 72 hours after dosing
  Residual area
Number of treatment-related adverse events (AE) for the test and the reference products as assessed by guidance predefined in the protocol | 28 days
  An AE is defined as any untoward medical occurrence in a subject administered an investigational product and which does not necessarily have a causal relationship with the treatment. The data from participants who had taken at least one investigational product was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Teteryukova, MD, Principal Investigator — National Anti-Doping Labaratory
Locations (1):
- National Anti-Doping Laboratory, Settl.Lesnoy, Minsk Oblast, Belarus

IPD SHARING:
Plan to Share IPD: Undecided
The Company may provide the individual participant data after privacy protection on the case by case basis